CLINICAL TRIAL: NCT05447741
Title: Fibromyalgia Versus Psoriatic Arthritis: Is Quantitative Ultrasound of the Enthesis a New Marker of Disease?
Brief Title: Quantitative Ultrasound of the Enthesis in Fibromyalgia and Psoriatic Arthritis
Status: Terminated | Type: Observational
Why Stopped: The recruitment and examination of participants were halted prematurely due to depleted funds.
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Other Study IDs: CE 21.405
Record Dates: First submitted 2022-06-08; First posted 2022-07-07 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia; Psoriatic Arthritis
MeSH Terms: conditions — Fibromyalgia; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with fibromyalgia: Participants will have a quantitative ultrasound examination of the dominant Achilles' tendon, medial collateral ligament at the femoral epicondyle and common extensor tendon at the lateral epicondyle of the elbow.
  Interventions: Diagnostic Test: Quantitative Ultrasound
- Patients with psoriasis arthritis: Participants will have a quantitative ultrasound examination of the dominant Achilles' tendon, medial collateral ligament at the femoral epicondyle and common extensor tendon at the lateral epicondyle of the elbow.
  Interventions: Diagnostic Test: Quantitative Ultrasound
- Asymptomatic controls: Participants will have a quantitative ultrasound examination of the dominant Achilles' tendon, medial collateral ligament at the femoral epicondyle and common extensor tendon at the lateral epicondyle of the elbow.
  Interventions: Diagnostic Test: Quantitative Ultrasound

INTERVENTIONS:
Diagnostic Test: Quantitative Ultrasound — Shear Wave Elastography acquisition. RF data acquisition (for HDK parameters calculation).

SUMMARY:
This prospective, cross-sectional, observational study will include subjects with fibromyalgia (FM), psoriatic arthritis (PsA) and asymptomatic controls. Participants will undergo a research ultrasound (US) exam of the enthesis of the Achilles' tendon, the medial collateral ligament at the femoral epicondyle and the common extensor tendon at lateral epicondyle of the elbow in resting conditions. The research US exam will consist of shear wave elastography (SWE) and radiofrequency (RF) data acquisitions. SWE technology will allow quantification of the shear wave speed (SWS) reporting the elastic stiffness of the tissues under investigation. RF data will be used to estimate quantitative ultrasound (QUS) parameters characterizing the mean intensity μ (akin to B-mode echogenicity), acoustic inhomogeneity (1/alpha), and structural spatial organization of echoes (κ) in the tissue.

DETAILED DESCRIPTION:
In this prospective, cross-sectional, observational study consecutive eligible subjects with FM, PsA, and a group of age- and sex-matched asymptomatic volunteers will undergo a research US examination of the dominant Achilles' tendon, knee medial collateral ligament and common extensor tendon of the elbow. Two operators under the supervision of a musculoskeletal radiologist will perform the US exam. B-mode and Power Doppler ultrasound of each tendon and ligament will be performed for morphological characterization. Then, shear wave elastography (SWE) and radiofrequency (RF) will be acquired. The shear wave speed (SWS) will be measured in the longitudinal plane using shear wave measurements. These features will be compared between groups. The HDK parameters (μ, 1/alpha, κ) will be computed offline, using RF sequences recorded in the longitudinal plane. Demographic features (participant age, sex, body mass index), the Leeds Enthesis Index (LEI) score assessed by the referring clinicians, and the self-administered Health Assessment Questionnaire (HAQ), Brief Pain Inventory (PBI) and Fibromyalgia Impact Questionnaire (FIQ) scores will be available for multivariate analyses.

ELIGIBILITY:
Inclusion Criteria Male and female subjects of all races and ethnic backgrounds aged between 18 - 60 years, able to provide informed consent and willing not to engage in sports activities for two days before the ultrasound (US) evaluation, will be considered eligible for this study.

Subjects with fibromyalgia:

* The diagnosis of fibromyalgia is based on the 2011 ACR criteria and confirmed by a pain medicine physician working at a tertiary care academic center (CHUM) having experience with patients with fibromyalgia and other chronic pain syndromes.
* Fibromyalgia is the primary reason for the patient's symptoms, without any other comorbid condition that could fully account for the symptoms of pain.
* No skin condition (psoriasis, eczema and others) requiring regular topical treatment.

Subjects with psoriatic arthritis:

* Presenting with psoriatic arthritis
* The diagnosis of psoriatic arthritis will be based on the ClASsification for Psoriatic Arthritis (CASPAR) criteria and established by a rheumatologist working at a tertiary care academic center (CHUM).
* No comorbid fibromyalgia as determined by the rheumatologist.

Asymptomatic subjects:

* No history of chronic pain syndromes, malformations, injuries, infections or tumors limiting activities of daily living and work.
* Not engaged in professional sports.
* No skin condition (psoriasis, eczema and others) requiring regular topical treatment.

Exclusion Criteria

* Pregnant and breast-feeding women
* History of spinal surgery or surgery to the extremities.
* Previous severe back or extremity fracture.
* Spinal or joint corticosteroid injections in the past 3 months.
* Major chronic illness (e.g., active cancer, inflammatory rheumatic disease other than psoriatic arthritis, or other chronic uncontrolled condition such as neurological, kidney, liver, cardiac, respiratory, or endocrine disease).
* Subjects unable to answer questionnaires in French or English.
* Subjects with psychiatric disorders that affect communication.
* Subjects who refused to participate.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with fibromyalgia will be recruited through various outreach approaches such as local newspapers, digital advertising on the Centre hospitalier de l'Université de Montréal (CHUM) platforms, and the collaboration of healthcare providers.
  Subjects with psoriatic arthritis will be recruited from those patients attending the rheumatology clinics at the CHUM.
  Asymptomatic volunteers will be recruited from the hospital community through local advertisements.
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-02-12 (Actual); Study Completion 2025-02-12 (Actual)

PRIMARY OUTCOMES:
Shear wave speed (SWS) (in m/sec). | Shear Wave Speed will be acquired when patients will be included in the study, from June 2022 to December 2023.
  Area under the ROC curve of the SWS to discriminate between groups.

SECONDARY OUTCOMES:
The quantitative ultrasound marker 'μ'. | The mean intensity μ will be acquired when patients will be included in the study, from June 2022 to December 2023.
  Statistical analysis of the echo envelope: the mean intensity μ. This marker is unitless.
  Area under the ROC curve of the μ parameter to discriminate between groups.
The quantitative ultrasound marker '1/alpha'. | the acoustic inhomogeneity 1/alpha parameter will be acquired when patients will be included in the study, from June 2022 to December 2023.
  Statistical analysis of the echo envelope: the acoustic inhomogeneity 1/alpha parameter. This marker is unitless.
  Area under the ROC curve of the 1/alpha parameter to discriminate between groups.
The quantitative ultrasound marker 'κ'. | The structure parameter κ will be acquired when patients will be included in the study, from June 2022 to December 2023.
  Statistical analysis of the echo envelope: the structure parameter κ. This marker is unitless.
  Area under the ROC curve of the κ parameter to discriminate between groups.
Inter-rater reliability | Shear Wave Elastography and RF data acquisitions that will be used for the inter-operator reliability measurements will be conducted when patients will be included in the study, from June 2022 to December 2023
  Estimation of the inter-operator reliability of the ultrasound parameter measurements on each enthesis.
  The inter-operator reliability will be assessed in terms of intraclass correlation coefficient (ICC 2,1) and coefficient of variation (CV).

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie J Bureau, MD MSc, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal, Montreal, Quebec, Canada